CLINICAL TRIAL: NCT03584243
Title: Evaluation of Efficiency and Security of Transepithelial Corneal Collagen Crosslinking With Oxygen to Treat Progressive Keratoconus.
Brief Title: Transepithelial Corneal Collagen Crosslinking in Eyes With Progressive Keratoconus
Acronym: TE-CXL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/17/0338; 2017-A02661-52 (Other: ID-RCB)
Record Dates: First submitted 2018-02-26; First posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Keratoconus
Keywords: collagen crosslinking; transepithelial crosslinking
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Intervention Model Description: This experimental study is a prospective, one-center city and non-comparative study.
  Patient with progressive keratoconus will be included after providing their consent. The intervention of the study is to perform transepithelial crosslinking with oxygen Outcomes will be evaluated from pretreatment baseline of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with progressive keratoconus (Experimental): Patient with progressive keratoconus will be included after providing their consent.
  The intervention administrated is a cross-linking with oxygen treatment
  Interventions: Procedure: A crosslinking with oxygen treatment

INTERVENTIONS:
Procedure: A crosslinking with oxygen treatment — A supplemental oxygen system during the cross linking will be used to apply filtered, humidified oxygen across the surface of the eye through a mask. The oxygen flow will be turned on immediately prior to initiation of irradiation, and will continue through the irradiation period. The supplemental oxygen flow will be shut off following completion of the programmed irradiation time.
  All subjects will be evaluated at screening, day 3, and 1, 3, 6, 12 and 24 months after treatment. At the same time all the potential adverse effects will be relieved.

SUMMARY:
Keratoconus is a corneal ectatic disease responsible for a loss of visual acuity when the steepening increases. Corneal collagen crosslinking (CXL) is a procedure that appears to halt or slow down the progression and avoid the visual impairment. However, such a technique requires the epithelium debridement, wich can be responsible for severs complications.

This study evaluate the safety and efficacy of transepithelial corneal crosslinking with oxygen to halt or slow down the progression of keratoconus. Such a procedure avoids the epithelium debridement and the related complications.

DETAILED DESCRIPTION:
Keratoconus is a common bilateral progressive corneal ectatic disease causing visual impairment by inducing irregular astigmatism and corneal opacities. This disorder typically begins during teenage years. Patients with severe forms may need a corneal transplantation. The CXL procedure, described in 1998, allows to halt or to slow down the disease progression and may avoid other surgeries, e.g. transplantation. This technique creates links between collagen fibrils in order to rigidify the corneal stroma. The corneal stroma is soaked with a riboflavin solution (vitamin B2) before being exposed to ultraviolet-A (UVA) radiations. In the current standard CXL, the central corneal epithelium must be debrided to allow the penetration of riboflavin into the cornea, with a risk of side effects, such as pain for the first two post-operative days, temporary loss of visual acuity during the first three months, and serious complications such as infections and stromal opacity due to corneal scarring Transepithelial crosslinking is a non-invasive technique in which benzalkonium chloride is used to enhance the penetration of riboflavin into the cornea. To improve the reaction, a device provides oxygen to the corneal surface. The transepithelial technique could allow intrastromal riboflavin diffusion, while keeping the corneal epithelium on, conserving the efficiency of the standard procedure without the complications induced by epithelial debridement.

Patient with progressive keratoconus will be included and treated with the transepithelial procedure. The follow-up will last for one year. Every follow-up visit will evaluate the security of the procedure and its efficacy to stop or slow down the progression of the disease. Interrogatory and slit lamp examination will be performed to investigate the potential adverse effects of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Provide written informed consent
* Diagnosis of progressive keratoconus
* Best corrected visual acuity between 0,05 and 1 decimal scale
* Willingness to follow all instructions and comply with schedule for follow-up visits.
* Social security insurance or equivalent.

Exclusion Criteria:

* Hypersensitivity to local treatment
* Corneal pachymetry < 400 μm
* Non progressive keratoconus
* Aphakic eye or eye with cataract implant without UV filter
* Concomitant corneal disease
* History of corneal surgery
* History of crosslinking treatment
* Pregnancy or lactation
* Juridical protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the transepithelial crosslinking method | One year
  The non-comparative evaluation of the efficacy of crosslinking of transepithelial corneal collagen with oxygen in the stabilization of progressive keratoconus during 12 months of follow-up.
  - Change from pretreatment baseline : keratometry at one year.
Efficacy of the transepithelial crosslinking method | One year
  The non-comparative evaluation of the efficacy of crosslinking of transepithelial corneal collagen with oxygen in the stabilization of progressive keratoconus during 12 months of follow-up.
  - Change from pretreatment in manifest refraction spherical equivalent at one year.
Efficacy of the transepithelial crosslinking method | One year
  - Change from pretreatment baseline : best corrected/uncorrected visual acuity at one year

SECONDARY OUTCOMES:
Security of the transepithelial crosslinking | One year
  The non-comparative evaluation of the safety of crosslinking of transepithelial corneal collagen with oxygen in the stabilization of progressive keratoconus during 12 months of follow-up.
  - Change from pretreatment baseline : intraocular pressure at one year.
Security of the transepithelial crosslinking | One year
  The non-comparative evaluation of the safety of crosslinking of transepithelial corneal collagen with oxygen in the stabilization of progressive keratoconus during 12 months of follow-up.
  - Change from baseline in endothelial cell count at one year.
Incidence and security of the transepithelial crosslinking | One year
  - Incidence of treatment emergent ocular adverse events reported during the study.
Incidence and security of the transepithelial crosslinking | One year
  - Percentage of eyes with loss in best corrected of three lines from pretreatment baseline.

CONTACTS AND LOCATIONS:
Overall Officials: François Malecaze, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No